CLINICAL TRIAL: NCT01301885
Title: Novel Diagnostic Tools for Endometriosis and Their Exploitation for Prognosis and Prevention of Complications
Brief Title: ENDOMET - Novel Diagnostic Tools and Treatments for Endometriosis
Acronym: ENDOMET
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government); VTT Technical Research Centre of Finland (Other); Finnish Medical Foundation (Network); Hormos Medical (Industry); PerkinElmer, Wallac Oy (Industry); Biotop Oy (Industry); Pharmatest Services Ltd (Unknown); Drug Discovery Graduate School, Finland (Unknown); The National Graduate School of Clinical Investigation, Finland (Unknown)
Responsible Party: Principal Investigator, Antti Perheentupa, Associate Professor, Turku University Hospital
Other Study IDs: ENDOMET-231/2004
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Endometriosis
Keywords: endometriosis; dysmenorrhea; infertility; biomarker; drug target; recurrence; complications; dyspareunia; dyschezia; dysuria; chronic pelvic pain; surgical treatment; long-term follow-up
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Infertility; Recurrence; Dyspareunia; Constipation; Dysuria | interventions — Laparoscopy; Laparotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, peritoneal fluid, endometrium tissue, healthy peritoneum, tissue of endometriosis (peritoneal, ovarian, deep infiltrating.
  Extracted DNA, RNA, cDNA and protein from the above samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endometriosis: Women (19-48 years of age) with surgically confirmed endometriosis.
  Interventions: Procedure: Laparoscopy/laparotomy
- Healthy women: Healthy women (32-48 years of age), symptom free, existence of endometriosis ruled out during laparoscopy for tubal ligation
  Interventions: Procedure: Laparoscopy/laparotomy

INTERVENTIONS:
Procedure: Laparoscopy/laparotomy — Surgical treatment of endometriosis (laparotomy/laparoscopy) or laparoscopic sterilisation. Sample collection in both groups.

SUMMARY:
Endometriosis is a chronic disease characterized by the presence of functional endometrial glands and stroma in ectopic locations outside the uterine cavity. The ectopic endometrial tissue responds to estradiol and other hormones similarly to the normal endometrium. Endometriosis is one of the most common benign gynecological conditions, as many as 5-10% of women in the reproductive age may be affected. In addition to pain which may be severe, subfertility is one of the typical problems associated with endometriosis and may be present in up to 40% of those affected. There is lack of a clear correlation between severity of pain and degree of compromised fertility. Different modes of treatment exist. Hormonal treatments are based on the suppression of estrogenic action on endometriosis as well as the endometrium. Unfortunately, discontinuation of the hormonal treatment typically results in a rapid recurrence of the disease. Surgery may alleviate the symptom for different lengths of time, however, curative treatment frequently involves hysterectomy with bilateral oophorectomy. In order to escape this radical treatment, new targeted therapy in the form of novel pharmacological agents would be of crucial importance. Presently, endometriosis can be reliably diagnosed only by laparoscopy. Since this is an invasive surgical procedure, new diagnostic tools would be warmly welcomed. Furthermore, as the progression of the disease is presently impossible to predict, new markers for the "malignancy" of each case are desperately needed.

The aim of the investigators research is to identify expression of endometriosis specific RNAs/proteins. Evaluation of expression profiles in samples of endometriosis and endometrium of patients with careful clinical and surgical classification of endometriosis as well as healthy control women should initially enable to identify novel targets for new therapies and biomarkers. Particularly the different pain symptoms will be recorded annually and evaluated comprehensively. Furthermore, combined with an adequate 10-year follow up (based on a questionnaire, including fertility, received treatments and different pain symptoms; NRS), the study should enable for example to identify markers for endometriosis associated infertility as well as cases where the disease progresses very rapidly or reoccurs. Different forms of effective treatment may thereafter be designed following the identification of such factors.

ELIGIBILITY:
Inclusion Criteria:

* study group: surgically and pathologically verified endometriosis
* control group: existence of endometriosis ruled out in laparoscopy

Exclusion Criteria:

* no other significant disease or medication for other diseases
* suspicion of malignancy
* pregnancy
* acute infection
* insufficient understanding of Finnish language
* previous hysterectomy and/or bilateral salpingo-oophorectomy

Ages: 19 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Endometriosis: Finnish Caucasian women surgically treated for endometriosis; age 19-48, no significant other disease or medication for other diseases
  Healthy controls: symptomless Finnish Caucasian women going through laparoscopy for tubal ligation; age 32-48, no significant other disease or medication
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2005-10; Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Intra-tissue steroid profiling indicates differential progesterone and testosterone metabolism in the endometrium and endometriosis lesions. | During the surgical sample collection
Endometrial and endometriotic concentrations of estrone and estradiol are determined by local metabolism rather than circulating levels. | During the surgical sample collection
Serum HE4 concentration differentiates malignant ovarian tumours from ovarian endometriotic cysts. | During the surgical sample collection
A relational database to identify differentially expressed genes in the endometrium and endometriosis lesions | During the surgical sample collection

SECONDARY OUTCOMES:
A prospective 5-year follow-up of pain recurrence after surgical treatment of endometriosis | 5 years (annually) after the completion of patient recruitment
  Questionnaire based evaluation of postoperative pain symptoms
Serum HE-4 concentration is not dependent on menstrual cycle or hormonal treatment among endometriosis patients and healthy premenopausal women | During surgical sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Antti Perheentupa, MD, PhD, Principal Investigator — Department of Obstetrics and Gynecology, Turku University Central Hospital
Locations (4):
- Finland (4):
  - Dept of Obstetrics and Gynecology, Helsinki University Hospital, Helsinki
  - Dept of Obstetrics and Gynecology, North Carelia Central Hospital, Joensuu
  - Dept of Obstetrics and Gynecology, Päijät-Häme Central Hospital, Lahti
  - Dept of Obstetrics and Gynecology, Turku University Central Hospital, Turku

REFERENCES:
- [Background] Gabriel M, Fey V, Heinosalo T, Adhikari P, Rytkonen K, Komulainen T, Huhtinen K, Laajala TD, Siitari H, Virkki A, Suvitie P, Kujari H, Aittokallio T, Perheentupa A, Poutanen M. A relational database to identify differentially expressed genes in the endometrium and endometriosis lesions. Sci Data. 2020 Aug 28;7(1):284. doi: 10.1038/s41597-020-00623-x. PMID 32859947
- [Background] Heinosalo T, Gabriel M, Kallio L, Adhikari P, Huhtinen K, Laajala TD, Kaikkonen E, Mehmood A, Suvitie P, Kujari H, Aittokallio T, Perheentupa A, Poutanen M. Secreted frizzled-related protein 2 (SFRP2) expression promotes lesion proliferation via canonical WNT signaling and indicates lesion borders in extraovarian endometriosis. Hum Reprod. 2018 May 1;33(5):817-831. doi: 10.1093/humrep/dey026. PMID 29462326
- [Result] Huhtinen K, Suvitie P, Hiissa J, Junnila J, Huvila J, Kujari H, Setala M, Harkki P, Jalkanen J, Fraser J, Makinen J, Auranen A, Poutanen M, Perheentupa A. Serum HE4 concentration differentiates malignant ovarian tumours from ovarian endometriotic cysts. Br J Cancer. 2009 Apr 21;100(8):1315-9. doi: 10.1038/sj.bjc.6605011. Epub 2009 Mar 31. PMID 19337252
- [Result] Hiissa J, Elo LL, Huhtinen K, Perheentupa A, Poutanen M, Aittokallio T. Resampling reveals sample-level differential expression in clinical genome-wide studies. OMICS. 2009 Oct;13(5):381-96. doi: 10.1089/omi.2009.0027. PMID 19663710
- [Result] Hallamaa M, Suvitie P, Huhtinen K, Matomaki J, Poutanen M, Perheentupa A. Serum HE4 concentration is not dependent on menstrual cycle or hormonal treatment among endometriosis patients and healthy premenopausal women. Gynecol Oncol. 2012 Jun;125(3):667-72. doi: 10.1016/j.ygyno.2012.03.011. Epub 2012 Mar 14. PMID 22426487
- [Result] Huhtinen K, Desai R, Stahle M, Salminen A, Handelsman DJ, Perheentupa A, Poutanen M. Endometrial and endometriotic concentrations of estrone and estradiol are determined by local metabolism rather than circulating levels. J Clin Endocrinol Metab. 2012 Nov;97(11):4228-35. doi: 10.1210/jc.2012-1154. Epub 2012 Sep 11. PMID 22969138
- [Result] Huhtinen K, Saloniemi-Heinonen T, Keski-Rahkonen P, Desai R, Laajala D, Stahle M, Hakkinen MR, Awosanya M, Suvitie P, Kujari H, Aittokallio T, Handelsman DJ, Auriola S, Perheentupa A, Poutanen M. Intra-tissue steroid profiling indicates differential progesterone and testosterone metabolism in the endometrium and endometriosis lesions. J Clin Endocrinol Metab. 2014 Nov;99(11):E2188-97. doi: 10.1210/jc.2014-1913. Epub 2014 Aug 19. PMID 25137424
- [Result] Vehmas AP, Muth-Pawlak D, Huhtinen K, Saloniemi-Heinonen T, Jaakkola K, Laajala TD, Kaprio H, Suvitie PA, Aittokallio T, Siitari H, Perheentupa A, Poutanen M, Corthals GL. Ovarian endometriosis signatures established through discovery and directed mass spectrometry analysis. J Proteome Res. 2014 Nov 7;13(11):4983-94. doi: 10.1021/pr500384n. Epub 2014 Aug 20. PMID 25099244